CLINICAL TRIAL: NCT00857818
Title: A 16-Week, Randomized, Controlled Trial of the Effect of Aripiprazole Versus Standard of Care on Non-HDL Cholesterol Among Patients With Schizophrenia and Bipolar I Disorder Who Have Pre-existing Metabolic Syndrome
Brief Title: Trial Comparing the Effects of Aripiprazole With Those of Standard of Care on Non-HDL Cholesterol in Patients With Schizophrenia or Bipolar I Disorder Who Have Metabolic Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN138-564
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2011-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar I Disorder; Metabolic Syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Metabolic Syndrome | interventions — Aripiprazole; Risperidone; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole (Experimental)
  Interventions: Drug: Aripiprazole
- Control group (Oanzapine, risperidone, or quetiapine) (Active Comparator)
  Interventions: Drug: Oanzapine, risperidone, or quetiapine

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole administered orally as tablets, 5 mg once daily (QD) in Week 1; 10 mg QD in Week 2. Flexible dosing allowed after Week 2, adjusted in 5-mg increments every 7 days within a range of 10 to 30 mg daily, for 16 weeks
  Other Names: Abilify; BMS-334039
  Arms: Aripiprazole
Drug: Oanzapine, risperidone, or quetiapine — Oanzapine, risperidone, or quetiapine administered orally as tablets at prior dosage for 16 weeks
  Arms: Control group (Oanzapine, risperidone, or quetiapine)

SUMMARY:
The purpose of this study was to determine whether patients with schizophrenia, schizoaffective disorder, or bipolar I disorder who also have metabolic syndrome have a larger decrease in fasting non-high density lipoprotein (non-HDL) cholesterol levels with aripiprazole than with their current atypical antipsychotic treatment (olanzapine, risperidone, or quetiapine).

ELIGIBILITY:
Inclusion Criteria:

* Competency in understanding nature of study and ability to sign informed consent form
* A clinical diagnosis of schizophrenia, schizoaffective disorder, or bipolar I disorder (manic or mixed) that has been treated with antipsychotics (oral olanzapine, risperidone or quetiapine) for at least 3 months.
* Treatment with any of the antipsychotic medications olanzapine, risperidone, or quetiapine for at least 3 months
* A Clinical Global Impression-Severity Scale score of 4 or lower at baseline
* Confirmed diagnosis of metabolic syndrome
* Patients not receiving treatment specifically for any of the parameters related to metabolic syndrome at the time of randomization
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and up to 4 weeks after last dose of investigational product
* Patients for whom it is clinically appropriate to switch from their current atypical antipsychotic to aripiprazole (determined by the investigator)

Exclusion Criteria:

* Risk of suicide (suicidal ideation or recently attempted suicide)
* Meeting Diagnostic and Statistical Manual of Mental Disorders, 4th ed, text revision criteria for any significant psychoactive substance use disorder within 3 months of screening
* Diagnosis of type 1 or 2 diabetes mellitus
* Current treatment for 1 of the components of metabolic syndrome
* Use of medication for the purpose of weight loss
* Diagnosis of bipolar disorders other than bipolar 1, depression with psychotic symptoms, or organic brain syndromes
* History of neuroleptic malignant syndrome
* Diagnosis of Parkinson's disease, Alzheimer's disease, multiple sclerosis, cerebral palsy, epilepsy, or mental retardation
* History of seizures
* Abnormal blood count for platelets, hemoglobin, absolute neutrophils, aspartate aminotransferase, alanine aminotransferase, creatinine, fasting glucose, and thyroid-stimulating hormone
* Electrocardiogram recording with QTc interval >475 msec
* Detectable levels of cocaine or positive screen for stimulants or other drugs considered (determined by the investigator) to be of abuse or dependence
* Blood alcohol levels superior or equal to 50 mg/dL [or 10.9 mmol/L]
* Prior participation in an aripiprazole clinical trial
* Treatment with aripiprazole within 1 month of enrollment
* Predefined exclusionary laboratory tests
* Patients with Bipolar Disorder treated with adjunctive therapy other than a stable dose of mood stabilizers (lithium or valproate) must undergo a 30-day washout period for adjunctive therapies, such as antidepressants, prior to randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- Canada (10):
  - Local Institution, Calgary, Alberta
  - Local Institution, Pentincton, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Hamilton, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Markham, Ontario
  - Local Institution, Mississauga, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 64 patients enrolled, 36 were screen failures, and 28 were randomized. Of those randomized, 26 received treatment.
Groups:
- Aripiprazole: 5 mg once daily (QD) in Week 1; 10 mg QD in Week 2. Flexible dosing allowed after Week 2, adjusted in 5-mg increments every 7 days in a range of 10 to 30 mg daily.
- Control Group (Olanzapine, Risperidone, or Quetiapine): Participants were to continue to receive the same dose of their current antipsychotic treatment (either olanzapine, risperidone, or quetiapine) for 16 weeks.
Period: Overall Study
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Started | 14 | 14
Received Treatment | 14 | 12
Completed | 3 | 6
Not Completed | 11 | 8
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Sponsor terminated study | 6 | 4
Not completed — Investigator decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine) | Total
Number analyzed (Participants) | 14 | 14 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 39.0 (10.36) | 32.9 (9.10) | 35.9 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 12 | 9 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Fasting Non-high Density Lipoprotein (Non-HDL) Cholesterol Levels
Description: Based on Last Observation Carried Forward data. Non-HDL cholesterol is defined as the difference between total cholesterol and high-density lipoprotein (HDL) cholesterol levels. Fasting non-HDL cholesterol is defined as the measured fasting HDL cholesterol level subtracted from the measured fasting total cholesterol level.
Time Frame: Baseline to Weeks 4, 8, and 16
Population: All randomized patients who took at least 1 dose of study medication during the treatment period. The Last Observation Carried Forward (LOCF) data set included data recorded at a given visit. If no observation was recorded at that visit, data was carried forward from the previous visit. .
Measure: Mean (Standard Error); unit: Percentage of change
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 13 | 12
Percentage of change
  Week 4 | -7.54 (3.22) | 0.19 (3.60)
  Week 8 | -18.45 (2.37) | -4.44 (2.86)
  Week 16 | -14.72 (3.86) | -2.47 (4.55)

2. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, and 1 or More AEs
Description: AE=any new untoward medical event or worsening of a preexisting medical condition that may or may not be causally related to treatment. SAE=any untoward medical occurrence that at any dose results in death; is life-threatening, a congenital anomaly/birth defect, or an important medical event; requires or prolongs inpatient hospitalization, or results in persistent or significant incapacity or drug dependency or abuse.
Time Frame: Baseline to Week 16, continuously
Population: All randomized subjects who took at least 1 dose of study medication during the treatment period.
Measure: Number; unit: Participants
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 14 | 14
Participants
  Deaths | 0 | 0
  SAEs | 2 | 0
  AEs leading to discontinuation | 3 | 0
  1 or more AEs | 11 | 6

3. Secondary Outcome: Mean Percent Changes From Baseline in Fasting Triglyceride and Total, High-Density Lipoprotein, and Low-Density Lipoprotein Cholesterol Levels
Time Frame: Baseline to Week 16
Population: Due to low enrollment, the study was terminated early. This endpoint was not analyzed because there were insufficient data to draw meaningful conclusions.
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Changes From Baseline in Fasting Glucose Levels
Time Frame: Baseline to Week 16
Population: as for outcome 3
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent of Participants Showing a Decrease or Increase in Body Weight of 7% or Greater From Baseline
Time Frame: Baseline and Weeks 4, 8, and 16
Population: as for outcome 3
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Changes From Baseline in Clinical Global Impression-Severity (CGI-S) Scale
Description: The CGI-S scale is a 7-point scale that requires the clinician to rate the severity of a patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; or 7=extremely ill.
Time Frame: Baseline and Weeks 4, 8, and 16
Population: as for outcome 3
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Changes From Baseline in Blood Pressure, Heart Rate, Hemoglobin Levels, White Blood Cell Count, Differential Count, and Absolute Platelet Count
Description: Any value falling outside of the normal range will be flagged for the attention of the investigator at the site. The investigator will indicate whether or not a flagged value is of clinical significance.
Time Frame: Baseline and Weeks 4, 8, and 16
Population: Due to low enrollment, this study was terminated early, and these data were not summarized.
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean Change From Baseline in Impact of Weight on Quality of Life (IWQoL-Lite) Scores
Description: The IWQoL-Lite is a 31-item self-report survey that assesses the impact of weight on quality of life (QoL) in obese patients. Total score=the sum of scores(ranging from 1-5 for each item) for all 31 items. The sum is then rescaled to a 0-100 scoring, with 0 representing the poorest and 100 the best QoL. The survey also assesses improvements in QoL that occur with weight losses of 5% or greater and deteriorations in QoL with weight gain of 5% or greater. A change of 7.8 to 12.0 points from baseline=meaningful improvement. A change of -4.5 to -7.6 points from baseline=meaningful deterioration.
Time Frame: Baseline to Weeks 4, 8, and 16
Population: as for outcome 3
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Mean Changes in Weight From Baseline
Time Frame: Baseline to Weeks 4, 8, and 16
Population: as for outcome 3
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Median Changes in Body Mass Index From Baseline
Time Frame: Baseline to Weeks 4, 8, and 16
Population: as for outcome 3
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Mean Changes in Serum Prolactin Levels From Baseline
Time Frame: Baseline to Weeks 4, 8. and 16
Population: as for outcome 3
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Mean Baseline Fasting Non-HDL Levels
Time Frame: At baseline (Day 1)
Population: All randomized patients who took at least 1 dose of study medication during the treatment period.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Aripiprazole | Control Group (Olanzapine, Risperidone, or Quetiapine)
Number analyzed (Participants) | 13 | 12
mg/dL | 176.07 (13.76) | 167.14 (14.01)

ADVERSE EVENTS:
Groups:
- CONTROL GROUP: Participants were to continue to receive the same dose of their current antipsychotic treatment (either olanzapine, risperidone, or quetiapine) for 16 weeks.
Arm/Group | ARIPIPRAZOLE | CONTROL GROUP
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/12
Other Adverse Events (participants affected / at risk) | 11/14 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARIPIPRAZOLE (N=14) | CONTROL GROUP (N=12)
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 | 0
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 | 0
PSYCHIATRIC DECOMPENSATION (Psychiatric disorders) | 1 | 0
NEUROLEPTIC MALIGNANT SYNDROME (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARIPIPRAZOLE (N=14) | CONTROL GROUP (N=12)
VISION BLURRED (Eye disorders) | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ANXIETY (Psychiatric disorders) | 2 | 0
INSOMNIA (Psychiatric disorders) | 3 | 0
AGITATION (Psychiatric disorders) | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 1 | 0
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 | 0
TREMOR (Nervous system disorders) | 3 | 0
HEADACHE (Nervous system disorders) | 1 | 0
AKATHISIA (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 1
PARAESTHESIA (Nervous system disorders) | 1 | 0
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
INCREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 1
FEELING HOT (General disorders) | 1 | 0
IRRITABILITY (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study terminated early due to low enrollment. Mean changes from baseline in: the Clinical Global Impression-Severity Scale and the Impact of Weight on Quality of Life scores were not analyzed due to insufficient data for meaningful conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.